CLINICAL TRIAL: NCT02186691
Title: Right and Left Ventricle Remodeling Predictors After Pulmonary Valve Replacement in Patients With Repaired Tetralogy of Fallot.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-06
Record Dates: First submitted 2014-06-04; First posted 2014-07-10 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Tetralogy of Fallot With Pulmonary Stenosis
Keywords: pulmonary valve replacement; tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RV and LV ejection fraction assesment (Experimental): assesment RV and LV ejection fraction after PVR measured by MRI
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI
  Other Names: assesment RV and LV ejection fraction after PVR

SUMMARY:
Long term survival of patients with repaired tetralogy of Fallot is excellent (about 85% at 35 year-old). However these patients are exposed to residual pulmonary stenosis (PS) and/or pulmonary regurgitation (PR). It is well established that these lesions can lead to irreversible sequelae such as right ventricle dilatation and dysfunction. Pulmonary valve replacement technique was developed to avoid long term right ventricular dysfunction. Pulmonary valve replacement indications are based upon the presence of symptoms at exercise and/or morphological or functional parameters such as severe pulmonary regurgitation with right ventricle dilatation/dysfunction. The best timing of such intervention is still underdebate with the main aim of having the right balance between avoiding long term sequelae of PR or PS and being the latter possible to push ahead the need for new intervention. Recent publication showed that myocardial diffuse fibrosis can contribute to irreversible alteration of myocardial contractility. Quantification of diffuse fibrosis by magnetic resonance imaging is feasible and could help the physician to best determine the right timing for PVR in this population of patients. Cardiac function assessment at rest and during exercise is possible using MR and our centre has developed a program for cardiac exercise during MRI. This could help to detect infra clinic abnormality and to analyse myocardial adaptation during exercise.

ELIGIBILITY:
Inclusion Criteria:

- older than 14 year-old, with repaired tetralogy of Fallot requiring pulmonary valve

Exclusion Criteria:

* liver failure, kidney failure,
* contra indication to MRI study,
* non-affiliated to the national health care program

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
determination of the quantity of diffuse myocardial fibrosis | 2.5 years
  determine if the quantity of diffuse myocardial fibrosis measured by cardiac magnetic resonnance (CMR) compare to baseline measure is correlated with decrease of RV volume and increase in RV and LV ejection fraction after PVR

SECONDARY OUTCOMES:
determination of contractile reserve | 2.5 years
  determine if contractile reserve measured by cardiac magnetic resonnance (CMR) compare to baseline measure is correlated with decrease of RV volume and increase in RV and LV ejection fraction after PVR

OTHER OUTCOMES:
determnation of variation fibrosis biomarkers | 2.5 years
  determine if the fibrosis biomarkers dosage compare to baseline measure is correlated with decrease of RV volume and increase in RV and LV ejection fraction after PVR

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice BONELLO, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France